CLINICAL TRIAL: NCT04470778
Title: A Phase 1, Open-label, Crossover Study to Assess the Effect of Acid-reducing Agent Famotidine on the Pharmacokinetics of BMS-986256 in Healthy Participants
Brief Title: Study to Assess the Effect of Acid-reducing Agent Famotidine on the Drug Levels of BMS-986256 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IM026-028
Record Dates: First submitted 2020-07-13; First posted 2020-07-14 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2022-11

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMS-986256 (Experimental)
  Interventions: Drug: BMS-986256
- BMS-986256 + Famotidine (Experimental)
  Interventions: Drug: BMS-986256; Drug: Famotidine

INTERVENTIONS:
Drug: BMS-986256 — Specified dose on specified days
Drug: Famotidine — Specified dose on specified days
  Arms: BMS-986256 + Famotidine

SUMMARY:
The purpose of this study is to investigate the effect of gastric pH changes due to famotidine administration on the drug levels of prototype BMS-986256 tablet formulation in healthy participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy participants having no clinically significant deviations from normal in medical history, physical examination (PE) findings, electrocardiograms (ECGs), vital signs, and clinical laboratory results that would compromise the ability to participate, complete, and/or interpret the results of the study
* Weight ≥ 50 kg and body mass index (BMI) between 18.0 kg/m2 and 32.0 kg/m2 inclusive at screening
* Women and men must agree to follow specific methods of contraception, if applicable, while participating in the trial

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Any significant acute or chronic medical illness
* Any major surgery within 4 weeks of study treatment administration
* Any other sound medical, psychiatric, and/or social reason as determined by the investigator

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2021-03-28 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 39 days
Area under the plasma concentration-time curve from time zero to time of the last quantifiable concentration AUC(0-T) | Up to 39 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time AUC(INF) | Up to 39 days

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 47 days
Incidence of Serious Adverse Events (SAEs) | Up to 74 days
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to 67 days
Incidence of clinically significant changes in clinical laboratory results: Clinical Chemistry tests | Up to 67 days
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | Up to 67 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 74 days
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 74 days
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 74 days
Incidence of clinically significant changes in vital signs: Heart rate | Up to 74 days
Incidence of clinically significant changes in 12-Lead electrocardiogram (ECG) parameters | Up to 74 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- ICON (LPRA) - Salt Lake, Salt Lake City, Utah, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm